CLINICAL TRIAL: NCT00035139
Title: Pediatric Traumatic Brain Injury: Methylphenidate Effects on Early Recovery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Murray Fellowship (Other)
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: NCRR-M01RR00240-1783
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Brain Injuries
Keywords: pediatric traumatic brain injury
MeSH Terms: conditions — Brain Injuries | interventions — Methylphenidate

INTERVENTIONS:
Drug: methylphenidate

SUMMARY:
Traumatic Brain Injury (TBI) is the leading cause of acquired long term disability among children and young adults. Deficits in attention and memory are common and persist for years after moderate or severe TBI. The similarity between these symptoms and those of children with AD/HD, the efficacy of methylphenidate in the treatment of AD/HD, and the efficacy of methylphenidate in improving recovery of animals with brain injuries, support the need to study methylphenidate effects in children with TBI. This investigation of methylphenidate in children with moderate to severe TBI aims to: (1) Assess the acute effects of 2 different dosages of methylphenidate on attention and reaction time when the medication is administered to children early in recovery; (2) Assess the ability of 8 weeks of methylphenidate to improve the rate of recovery of cognitive, memory, and attentional skills in children with TBI; (3) Identify the frequency of common methylphenidate side effects in children with TBI.

DETAILED DESCRIPTION:
During the first phase of the study which is of 8-days duration subjects will receive placebo on some days and methylphenidate on others. During this phase of the study the effects of the medication on children's performance on a computerized test of attention will be assessed. Individuals who do not have significant methylphenidate side effects during the first phase of the study will then participate in the second phase of the study. During the second phase subjects will receive either methylphenidate or placebo for 8 weeks. Neuropsychological measures of attention, memory, behavioral inhibition, cognitive flexibility, and motor performance will be obtained at baseline and after the 8 week medication trial in order to assess methylphenidate effects on the rate of recovery. Recovery will also be assessed using an interview measure of adaptive behavior and cognitive functioning. A stimulant medication side effect rating scale will be used to monitor for common methylphenidate adverse effects throughout both phases of the study

ELIGIBILITY:
Moderate to severe traumatic brain injury

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child

CONTACTS AND LOCATIONS:
Locations (1):
- Childrens Hospital Of Philadelphia, Philadelphia, Pennsylvania, United States